CLINICAL TRIAL: NCT00763958
Title: Relapse Prevention to Reduce HIV Among Women Prisoners
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karen Cropsey, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R21DA019838 (NIH); 5R21DA019838-03 (NIH); 7R21DA019838-02 (NIH)
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Results first posted 2012-06-04 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Opioid Dependence; HIV
Keywords: opiates; HIV
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine (Experimental): Active sublingual buprenorphine provided to participants; dose as clinically indicated up to 32 mg daily for up to 3 months
  Interventions: Drug: Buprenorphine
- Placebo (Placebo Comparator): Placebo sublingual medication provided to individuals randomized to control up to 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to match buprenorphine administered for 3 months
  Arms: Placebo
Drug: Buprenorphine — Buprenorphine provided for 3 months; dosing was as clinically indicated up to 32 mg daily.
  Arms: Buprenorphine

SUMMARY:
This study is a feasibility and acceptability study assessing whether providing buprenorphine for women under criminal justice supervision leaving a controlled environment and returning to the community would prevent opioid relapse and reduce HIV risk behaviors.

DETAILED DESCRIPTION:
This study sought to enroll opioid dependent women under supervision in the criminal justice system and in a controlled environment (substance abuse treatment)but at at high risk for opioid relapse and engaging in HIV risk behaviors when returning to the community. Initially, 9 women were enrolled and received buprenorphine medication. After the first 9 participants, women were randomized to either buprenorphine or placebo. Women received the buprenorphine medication for 12 weeks in the community and at the end of the 12 weeks were transitioned either to another buprenorphine provider, methadone provider, or tapered off buprenorphine based on the participant's preferences. One additional follow-up at 3 months after treatment was conducted. The primary outcome was opioid positive urines at all time points.

ELIGIBILITY:
Inclusion Criteria:

* female,
* history of opioid dependence,
* released back to the community from a controlled environment,
* criminal justice involvement.

Exclusion Criteria:

* under age 19,
* medical contraindications,
* major psychiatric problems.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in May of 2008 and ended June of 2010. All participants were recruited from a 28-day drug inpatient facility that accepts patients from the criminal justice system.
Pre-assignment Details: Initially, 11 women were enrolled in the open-label trial, followed by 33 women randomized to either buprenorphine or placebo.
Groups:
- Buprenorphine: Buprenorphine provided for 12 weeks up to 32 mg daily based on clinical assessment.
- Placebo: Medication "sugar pill" provided for 12 weeks up to 32 mg daily.
Period: Overall Study
Arm/Group | Buprenorphine | Placebo
Started | 28 | 16
Completed | 14 | 5
Not Completed | 14 | 11
Not completed — did not meet final criteria | 4 | 4
Not completed — Lost to Follow-up | 10 | 2
Not completed — Believed they were receiving placebo | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine | Placebo | Total
Number analyzed (Participants) | 28 | 16 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 16 | 44
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.2 (6.6) | 34.7 (10.3) | 31.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 44
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Opiate Positive Urines With Missing Urines Coded as Positive at Week 12.
Description: Number of participants with positive opiate urine samples at 12 weeks of treatment.
Time Frame: 12 weeks
Population: All subjects were included in the analysis population as intent to treat.
Measure: Number; unit: participants
Groups:
- Buprenorphine: Buprenorphine provided for 12 weeks of study drug based on clinical assessment.
- Placebo: Medication "sugar pill" provided for 12 weeks.
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 24 | 12
participants | 14 | 5

2. Secondary Outcome: Number of Participants Who Enroll in the Study.
Description: To determine the number of participants who enroll in the study during the time of recruitment.
Time Frame: up to 24 months
Measure: Number; unit: participants
Groups:
- Buprenorphine: Buprenorphine provided for 12 weeks of stuty drug based on clinical assessment.
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 28 | 16
participants | 28 | 16

3. Primary Outcome: Opiate Positive Urines With Missing Urines Coded as Positive at Week 24.
Description: Number of participants with positive opiate urine sample at the 24 week follow-up.
Time Frame: 24 weeks
Population: All subjects were included in the analysis population as intent to treat.
Measure: Number; unit: participants
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 24 | 12
participants | 4 | 4

ADVERSE EVENTS:
Arm/Group | Buprenorphine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/16
Other Adverse Events (participants affected / at risk) | 0/28 | 0/16

LIMITATIONS AND CAVEATS:
Slow recruitment with poor retention. Transient population that was difficult to effectively track.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No